CLINICAL TRIAL: NCT03160144
Title: Effects of Open Lung Approach on Intraoperative Respiratory Function and Postoperative Recovery of Patients With Laparoscopic Colorectal Resection
Brief Title: The PROtective Ventilation Using Open Lung Approach Or Not Trial
Acronym: PROVOLON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hong Li, Principal Investigator, The department of anesthesiology, Sixth Affiliated Hospital, Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017ZSLYEC-002
Record Dates: First submitted 2017-04-21; First posted 2017-05-19 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Pulmonary Complications; Respiratory Insufficiency
Keywords: laparoscopic resection of colorectal cancer; open lung approach
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open lung approach ventilation strategy (Experimental): Procedure: open lung approach ventilation strategy (OLV). Patients receive volume-controlled mechanical ventilation with a tidal volume of 6 to 8 ml per kilogram of predicted body weight, a PEEP of 6 to 8 cm of water, and recruitment maneuvers repeated every 30 minutes after tracheal intubation.
  Interventions: Procedure: open lung approach
- conventional ventilation strategy (No Intervention): Procedure: conventional ventilation strategy (NOLV). Patients receive volume-controlled mechanical ventilation with a tidal volume of 6 to 8 ml per kilogram of predicted body weight, no PEEP and no recruitment maneuver.

INTERVENTIONS:
Procedure: open lung approach
  Other Names: open lung strategy
  Arms: open lung approach ventilation strategy

SUMMARY:
Postoperative Pulmonary Complications (PPC) are very common. It severely affects postoperative recovery, particularly in the abdominal surgery. Patients with laparoscopic resection of colorectal cancer generally have a higher age and decreased lung function reserve. At the same time, they prone to developing atelectasis due to the effects of pneumoperitoneum pressure. Therefore, they are a high-risk group of respiratory insufficiency and PPC.

Mechanical ventilation with a low tidal volume is a routine in clinic nowadays. However, this conventional strategy will also result in atelectasis formation. Therefore, it may deteriorate the vulnerable lung function of patients undergoing laparoscopic resection of colorectal cancer. Patients with Acute Lung Injury or Acute Respiratory Distress Syndrome (ALI/ARDS) could benefit from the "open lung approach", including the use of positive end-expiratory pressure (PEEP) and recruitment maneuvers (RMs). Whether a lung protective mechanical ventilation strategy with medium levels of PEEP and repeated RMs, the "open lung approach", protects against respiratory insufficiency and PPC during laparoscopic resection of colorectal cancer is uncertain. The present study aims at comparing the effects of "open lung approach" mechanical ventilation strategy and conventional mechanical ventilation strategy in PPC, extra-pulmonary complications, length of hospital stay, biomarkers of lung injury and changes of respiratory function in patients undergoing general anesthesia for laparoscopic resection of colorectal cancer.

DETAILED DESCRIPTION:
1. Sample size calculation, randomization and patients safety. The required sample size is calculated from previous studies on the incidence of postoperative pulmonary complications. A two group chi-square test with a 0.05 two-sided significance level will have 80% power to detect the difference (in primary outcome) between conventional mechanical ventilation strategy (25%) and open lung approach mechanical ventilation strategy (12.5%) when the sample size in each group is 126. In consideration of a 10% loss rate, 280 cases to be included in this trial.

   Research will be carried out in two stages. Completely-randomized design was used in the first stage, and randomized block design in the second stage. The interim analysis will be performed when 100 patients (first stage) have successfully been included and followed-up. The Data Monitoring and Safety Group (DMSG) will provide recommendations about stopping or continuing the trial to the principal investigator. The DMSG will recommend stopping the trial, if significant group-difference in adverse events is found at the interim analysis (p<0.025), or if postoperative pulmonary complications occur more frequently in the intervention group (p<0.025). If the intervention has a strong trend for improving postoperative pulmonary complications (p<0.018) at the first stage, termination of the study is considered.
2. Protocol drop-out. Anesthesiologists are allowed to change the ventilation protocol if there is any concern about patient's safety. The level of PEEP can be modified according to the anesthesiologist in charge if the systolic arterial pressure (SBP)< 80 mmHg and SBP drop ≥30% baseline values for more than 3 minutes despite intravenous fluid infusion and/or start of vasopressors, if dosages of vasopressors are at the highest level tolerated, if new arrhythmias develop which are unresponsive to treatment suggested by the Advanced Cardiac Life Support Guidelines. If there is pneumothorax or hypoxemia (SpO2 < 90% for more than 3 minutes）, if there is need of massive transfusion (>8 units packed red blood cell) to maintain hemoglobin >7 mg/dl, if the duration of pneumoperitoneum is less then 1h or mechanical ventilation time is less then 2h, if there is a surgical complication (such as severe hypercapnia, unexpected conversion to open surgery, unplanned reoperation in 24h after surgery, unplanned ICU admission for surgical reasons) or if patient die during operation, then the patient will be dropped out of the study. All drop-out cases will be included in the safety analysis.
3. Trial settings for intraoperative ventilation. Patients in the conventional mechanical ventilation strategy group will have a tidal volume of 6 to 8 ml per kilogram Predicted Body Weight (PBW), zero PEEP and no recruitment maneuver. Patients in the open lung approach mechanical ventilation strategy group will have a tidal volume of 6 to 8 ml per kilogram PBW, a PEEP level of 6 to 8 cm of water and recruitment maneuvers. Recruitment maneuvers consist of a stepwise increase of tidal volume （as detailed below） and will be applied immediately after tracheal intubation and every 30 min thereafter until the end of surgery.

   In each group, anesthesiologists will be advised to use an inspired oxygen fraction (FIO2) between 0.4 to 0.5 and to maintain oxygen saturation ≥ 92%. The inspiratory to expiratory time ratio will be set at 1:2, with a respiratory rate adjusted to maintain normocapnia (end-tidal carbon dioxide concentration of 30-50 mmHg).

   PBW is calculated according to a predefined formula with: 50 + 0.91 x (centimeters of height - 152.4) for males and 45.5 + 0.91 x (centimeters of height - 152.4) for females. In each group, patients will be ventilated using the volume-controlled ventilation strategy using an anesthesia ventilator: 1. Avance® (Datex-Ohmeda, General Electric, Helsinki, Finland) 2. Tiro® (Dräger, Lübeck, Germany)
4. Recruitment maneuvers.

   Stepwise increase of tidal volume will be used as a method of recruitment maneuvers in this trial. Recruitment maneuvers should not be performed when patients are hemodynamic unstable, as judged by the attending anesthesiologist. Recruitment maneuvers will be performed as follows:

   4-1. Peak inspiratory pressure limit is set at 45 cmH2O. 4-2. Tidal volume is set at 8 ml/kg PBW and respiratory rate at 6 breaths/min, while PEEP is set at 12 cmH2O.

   4-3. Inspiratory to expiratory ratio (I:E) is set at 1:2. 4-4. Tidal volumes are increased in steps of 4 ml/kg PBW until a plateau pressure of 30-35 cmH2O (if tidal volume reach the biggest volume of the ventilator and plateau pressure cannot reach 30-35 cmH2O, then PEEP is set at 16 cmH2O for a plateau pressure of 30-35 cmH2O).

   4-5. Three breaths are administered with a plateau pressure of 30-35 cmH2O. 4-6. Peak inspiratory pressure limit, respiratory rate, I: E, and tidal volume are set back to settings preceding each recruitment maneuver, while maintaining PEEP at 8 cmH2O.
5. Definitions for postoperative complications. All definitions for postoperative complications refer to the IMPROVE trial and the PROVHILO trial.
6. Composition and responsibilities of the DMSG. Members of the DMSG are the management team of anesthesia department in the research hospital. The DMSG will be responsible for safeguarding the interests of trial participants, assessing the safety and efficacy of the intervention during the trial, and for monitoring the overall conduct of the trial. To enhance the integrity of the trial, the DMSG may also formulate recommendations relating to the selection or recruitment of participants, and the procedures of data management and quality control. The DMSG will be advisory to the principal investigator. The principal investigator will be responsible for reviewing the DMSG recommendations, decide whether to continue or terminate the trial, and determine whether changes in trial conduct are required. Any DMSG members who develop significant conflicts of interest during the course of the trial should resign from the DMSG.
7. Data management. Data will be collected and recorded into case report forms (CRFs) by researchers under the supervision of DMSG members. Data manager will scan handwritten data first and then enter data into electronic database. Source data verification will be performed using a cross-check method by researchers when 7-days follow-up have successfully been completed.

   All adverse events, serious adverse events, unexpected or possibly related events will be recorded in the CRF and reported to the DMSG.
8. Statistics. Statisticians will be in blind state for data analysis. Analysis will be by intention-to-treat comparing the primary outcome measure at 7 days in the two groups by chi-squared test (or Fisher's exact test as appropriate). Continuous variables will be compared using the One-way analysis of variance or the Mann-Whitney U test. Categorical variables will be compared using the chi-square test or the Fisher's exact test. The time-to-event curves will be calculated with the use of the Kaplan-Meier method. All analyses will be conducted using the SPSS 16.0 statistical software.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years.
2. Undergo elective laparoscopic resection of colorectal cancer.
3. With an expected duration of pneumoperitoneum ≥1.5h.
4. With a preoperative risk index for pulmonary complications ≥ 2.
5. With no contraindication of epidural anesthesia.
6. Pulse oxygen saturation in air ≥ 92%.
7. And informed consent obtained.

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status ≥ IV.
2. Body mass index ≥30kg/m2.
3. Duration of mechanical ventilation ≥ 1h within 2 weeks preceding surgery.
4. A history of acute respiratory failure within 1 month preceding surgery.
5. With a sepsis or septic shock or instable hemodynamics.
6. With a progressive neuromuscular illness such as myasthenia gravis.
7. With a epilepsy or schizophrenia or Parkinson's disease.
8. With a severe chronic obstructive pulmonary disease (COPD) or pulmonary bulla.
9. Severe organ dysfunction (acute coronary syndrome, uremia, hepatic encephalopathy, classification of function capacity of the NYHA ≥III, malignant arrhythmia and so on).
10. Coma, severe cognitive deficit, language or hearing impairment who cannot communicate.
11. Not proper controlled hypertension.
12. Involved in other clinical studies or refused to join in the research.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Occurrence rate of major pulmonary and extrapulmonary complications | Day 0 to 7 after surgery
  Major pulmonary complications were defined as suspected pneumonia，acute respiratory failure and sustained hypoxia; Major extrapulmonary complications were defined as sepsis, severe sepsis and septic shock or death.

SECONDARY OUTCOMES:
Peak airway Pressure | Intraoperative, period of mechanical ventilation
  Peak airway Pressure（Ppeak, cm H2O);
Plateau airway pressure | Intraoperative, period of mechanical ventilation
  Plateau airway pressure（Pplat, cm H2O）;
Static lung compliance | Intraoperative, period of mechanical ventilation
  Static lung compliance (Csta, ml/cm H2O) = Vt/ (Pplat-PEEP);
Dynamic lung compliance | Intraoperative, period of mechanical ventilation
  Dynamic lung compliance (Cdyn , ml/cm H2O)= Vt/ (Ppeak-PEEP);
Arterial partial pressure of oxygen | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Arterial partial pressure of oxygen (PaO2, mmHg）; post-anaesthesia care unit (PACU);
Alveolar-arterial oxygen tension difference | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Alveolar-arterial oxygen tension difference (A-aDO2, mmHg）;
Arterial- alveolar oxygen tension ratio | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Alveolar oxygen pressure (PAO2); Arterial- alveolar oxygen tension ratio ( a / A ratio) =PaO2 / PAO2;
Respiratory index | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Fraction of inspired oxygen (FiO2); Respiratory index (RI) = P(A-a)DO2/ FiO2;
Oxygenation index | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Oxygenation index (OI)=PaO2/FiO2;
Alveolar dead space fraction | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Arterial carbon dioxide partial pressure (PaCO2); partial pressure of carbon dioxide in endexpiratory gas (PetCO2); Alveolar dead space fraction (Vd/Vt）=(PaCO2-PetCO2)/ PaCO2;
Lactic acid | pre-anesthesia, 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Lactic acid ( LAC, mmol/L);
Oxygen extraction ratio | The first stage of the study: 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Oxygen content of central venous blood (CvO2); Oxygen content of arterial blood (CaO2); oxygen extraction ratio (O2ER)＝(CaO2-CvO2) /CaO2;
Central venous blood oxygen saturation | The first stage of the study: 0.5 hour after pneumoperitoneum, 1.5 hours after pneumoperitoneum, 20 minutes after entering PACU
  Central venous blood oxygen saturation (ScvO2).
Advanced glycation end products receptor | Intraoperative (pre-anesthesia, post-operation) and postoperative (postoperative day 3)
  Advanced glycation end products receptor (RAGE, pg/ml).
S100 beta protein | Intraoperative (pre-anesthesia, post-operation) and postoperative (postoperative day 3)
  S100 beta protein （S100β, μg/L）.
Tumor Necrosis Factor alpha | Intraoperative (pre-anesthesia, post-operation) and postoperative (postoperative day 3)
  Tumor Necrosis Factor alpha (TNF-α, pg/ml);
Interleukin 6 | Intraoperative (pre-anesthesia, post-operation) and postoperative (postoperative day 3)
  Interleukin 6 (IL-6, pg/ml).
The occurrence rate of hypoxemia in PACU | 20 minutes after entering PACU
  The occurrence rate of hypoxemia (PaO2<60 mmhg) in PACU
Length of PACU stay | Though study completion, an average of half an hour.
  Length of PACU stay (min);
The recovery time from anesthesia | Though study completion, an average of one hour.
  The recovery time from anesthesia (min).
Postoperative pulmonary complications | Day 0 to 7 after surgery
  The incidence of postoperative pulmonary complications based on a PPC scale.
Postoperative acute respiratory failure | Day 0 to 7 after surgery
  Occurrence rate of acute respiratory failure (SpO2< 90% or PaO2<60mmhg);
Postoperative suspected pneumonia | Day 0 to 7 after surgery
  Occurrence rate of postoperative pneumonia;
Pulse oximetry less than 92% | Day 0 to 7 after surgery
  Occurrence rate of saturation of pulse oximetry less than 92%;
Sustained hypoxia | Day 0 to 7 after surgery
  Occurrence rate of sustained hypoxia
Saturation of pulse oximetry | Day 0 to 7 after surgery
  Saturation of pulse oximetry (SpO2);
Occurrence rate of intervention-related adverse events | Intraoperative, period of mechanical ventilation
  Intervention-related adverse events including: rescue therapy for desaturation, potentially harmful hypotension, pneumothorax, vasoactive drugs needed.
Postoperative delirium | Day 1 to 3 after surgery
  Postoperative delirium will be estimated by a scale called Confusion Assessment Method-ICU.
Occurrence rate of related complications | Day 0 to 7 after surgery
  Related complications including: the systemic inflammatory response syndrome (SIRS), acute myocardial infarction (AMI), Acute hepatic and renal insufficiency; surgical complications including intraabdominal abscess, anastomotic leakage.
Unplanned reoperation after 24h | Up to 30 days after surgery
  Unplanned reoperation after 24h (operation not caused by bleeding in 24h).
Postoperative hospital stay | Up to 30 days after surgery
  Postoperative hospital stay.
Lung recruitment maneuver systolic blood pressure changes | The first stage of the study: intraoperative, when lung recruitment maneuver is operated.
  Systolic blood pressure (SBP, mmHg);
Lung recruitment maneuver related diastolic blood pressure changes | The first stage of the study: intraoperative, when lung recruitment maneuver is operated.
  Diastolic blood pressure (DBP, mmHg);
Lung recruitment maneuver related mean arterial pressure changes | The first stage of the study: intraoperative, when lung recruitment maneuver is operated.
  Mean arterial pressure (MBP, mmHg); heart rate (HR, bpm).
Lung recruitment maneuver related heart rate changes | The first stage of the study: intraoperative, when lung recruitment maneuver is operated.
  Heart rate (HR, bpm).
Death from any cause. | Up to 30 days after surgery
  Death from any cause 30 days after surgery.
Unplanned admission to ICU | Up to 30 days after surgery
  Unplanned admission to ICU (not caused by bleeding in 24h).
Impaired oxygenation | before anesthesia induction, 0.5 h and 1.5 h after pneumoperitoneum induction, and 20 min after postanesthesia care unit (PACU) admission
  PaO2/FIO2 ≤ 300 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University; Hong Li, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The sixth affiliated hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Smetana GW. Preoperative pulmonary evaluation. N Engl J Med. 1999 Mar 25;340(12):937-44. doi: 10.1056/NEJM199903253401207. No abstract available. PMID 10089188
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Brooks-Brunn JA. Predictors of postoperative pulmonary complications following abdominal surgery. Chest. 1997 Mar;111(3):564-71. doi: 10.1378/chest.111.3.564. PMID 9118688
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Gajic O, Dara SI, Mendez JL, Adesanya AO, Festic E, Caples SM, Rana R, St Sauver JL, Lymp JF, Afessa B, Hubmayr RD. Ventilator-associated lung injury in patients without acute lung injury at the onset of mechanical ventilation. Crit Care Med. 2004 Sep;32(9):1817-24. doi: 10.1097/01.ccm.0000133019.52531.30. PMID 15343007
- [Background] Lee WL, Detsky AS, Stewart TE. Lung-protective mechanical ventilation strategies in ARDS. Intensive Care Med. 2000 Aug;26(8):1151-5. doi: 10.1007/s001340051332. No abstract available. PMID 11030175
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Wanderer JP, Blum JM, Ehrenfeld JM. Intraoperative low-tidal-volume ventilation. N Engl J Med. 2013 Nov 7;369(19):1861. doi: 10.1056/NEJMc1311316. No abstract available. PMID 24195560
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Guay J, Ochroch EA. Intraoperative use of low volume ventilation to decrease postoperative mortality, mechanical ventilation, lengths of stay and lung injury in patients without acute lung injury. Cochrane Database Syst Rev. 2015 Dec 7;(12):CD011151. doi: 10.1002/14651858.CD011151.pub2. PMID 26641378
- [Background] Cox PN, Bryan AC. Small tidal volumes and the open-lung approach. Crit Care Med. 2001 Apr;29(4):915. doi: 10.1097/00003246-200104000-00056. No abstract available. PMID 11373501
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Hedenstierna G. Re-expansion of atelectasis during general anaesthesia: a computed tomography study. Br J Anaesth. 1993 Dec;71(6):788-95. doi: 10.1093/bja/71.6.788. PMID 8280539
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Jaber S, Coisel Y, Chanques G, Futier E, Constantin JM, Michelet P, Beaussier M, Lefrant JY, Allaouchiche B, Capdevila X, Marret E. A multicentre observational study of intra-operative ventilatory management during general anaesthesia: tidal volumes and relation to body weight. Anaesthesia. 2012 Sep;67(9):999-1008. doi: 10.1111/j.1365-2044.2012.07218.x. Epub 2012 Jun 18. PMID 22708696
- [Background] Hess DR, Kondili D, Burns E, Bittner EA, Schmidt UH. A 5-year observational study of lung-protective ventilation in the operating room: a single-center experience. J Crit Care. 2013 Aug;28(4):533.e9-15. doi: 10.1016/j.jcrc.2012.11.014. Epub 2013 Jan 29. PMID 23369521
- [Background] Levin MA, McCormick PJ, Lin HM, Hosseinian L, Fischer GW. Low intraoperative tidal volume ventilation with minimal PEEP is associated with increased mortality. Br J Anaesth. 2014 Jul;113(1):97-108. doi: 10.1093/bja/aeu054. Epub 2014 Mar 12. PMID 24623057
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Reber A, Hedenstierna G. Prevention of atelectasis during general anaesthesia. Lancet. 1995 Jun 3;345(8962):1387-91. doi: 10.1016/s0140-6736(95)92595-3. PMID 7760608
- [Background] Takahata O, Kunisawa T, Nagashima M, Mamiya K, Sakurai K, Fujita S, Fujimoto K, Iwasaki H. Effect of age on pulmonary gas exchange during laparoscopy in the Trendelenburg lithotomy position. Acta Anaesthesiol Scand. 2007 Jul;51(6):687-92. doi: 10.1111/j.1399-6576.2007.01311.x. Epub 2007 Apr 26. PMID 17465975
- [Background] Retamal J, Borges JB, Bruhn A, Cao X, Feinstein R, Hedenstierna G, Johansson S, Suarez-Sipmann F, Larsson A. High respiratory rate is associated with early reduction of lung edema clearance in an experimental model of ARDS. Acta Anaesthesiol Scand. 2016 Jan;60(1):79-92. doi: 10.1111/aas.12596. Epub 2015 Aug 10. PMID 26256848
- [Background] Duggan M, Kavanagh BP. Pulmonary atelectasis: a pathogenic perioperative entity. Anesthesiology. 2005 Apr;102(4):838-54. doi: 10.1097/00000542-200504000-00021. PMID 15791115
- [Background] Arozullah AM, Khuri SF, Henderson WG, Daley J; Participants in the National Veterans Affairs Surgical Quality Improvement Program. Development and validation of a multifactorial risk index for predicting postoperative pneumonia after major noncardiac surgery. Ann Intern Med. 2001 Nov 20;135(10):847-57. doi: 10.7326/0003-4819-135-10-200111200-00005. PMID 11712875
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Guldner A, Kiss T, Serpa Neto A, Hemmes SN, Canet J, Spieth PM, Rocco PR, Schultz MJ, Pelosi P, Gama de Abreu M. Intraoperative protective mechanical ventilation for prevention of postoperative pulmonary complications: a comprehensive review of the role of tidal volume, positive end-expiratory pressure, and lung recruitment maneuvers. Anesthesiology. 2015 Sep;123(3):692-713. doi: 10.1097/ALN.0000000000000754. PMID 26120769
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Citerio G, Pesenti A, Latini R, Masson S, Barlera S, Gaspari F, Franzosi MG; NeuroMorfeo Study Group. A multicentre, randomised, open-label, controlled trial evaluating equivalence of inhalational and intravenous anaesthesia during elective craniotomy. Eur J Anaesthesiol. 2012 Aug;29(8):371-9. doi: 10.1097/EJA.0b013e32835422db. PMID 22569025
- [Background] Hemmes SN, Severgnini P, Jaber S, Canet J, Wrigge H, Hiesmayr M, Tschernko EM, Hollmann MW, Binnekade JM, Hedenstierna G, Putensen C, de Abreu MG, Pelosi P, Schultz MJ. Rationale and study design of PROVHILO - a worldwide multicenter randomized controlled trial on protective ventilation during general anesthesia for open abdominal surgery. Trials. 2011 May 6;12:111. doi: 10.1186/1745-6215-12-111. PMID 21548927
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Jiang SP, Li ZY, Huang LW, Zhang W, Lu ZQ, Zheng ZY. Multivariate analysis of the risk for pulmonary complication after gastrointestinal surgery. World J Gastroenterol. 2005 Jun 28;11(24):3735-41. doi: 10.3748/wjg.v11.i24.3735. PMID 15968730
- [Background] Xu T, Bo L, Wang J, Zhao Z, Xu Z, Deng X, Zhu W. Risk factors for early postoperative cognitive dysfunction after non-coronary bypass surgery in Chinese population. J Cardiothorac Surg. 2013 Nov 1;8:204. doi: 10.1186/1749-8090-8-204. PMID 24175992
- [Background] Jabaudon M, Futier E, Roszyk L, Sapin V, Pereira B, Constantin JM. Association between intraoperative ventilator settings and plasma levels of soluble receptor for advanced glycation end-products in patients without pre-existing lung injury. Respirology. 2015 Oct;20(7):1131-8. doi: 10.1111/resp.12583. Epub 2015 Jun 29. PMID 26122046
- [Derived] Li H, Luo TF, Zhang NR, Zhang LZ, Huang X, Jin SQ. Factors associated with prolonged postoperative length of hospital stay after laparoscopic colorectal cancer resection: a secondary analysis of a randomized controlled trial. BMC Surg. 2022 Dec 24;22(1):438. doi: 10.1186/s12893-022-01886-4. PMID 36566186
- [Derived] Li H, Zheng ZN, Zhang NR, Guo J, Wang K, Wang W, Li LG, Jin J, Tang J, Liao YJ, Jin SQ. Intra-operative open-lung ventilatory strategy reduces postoperative complications after laparoscopic colorectal cancer resection: A randomised controlled trial. Eur J Anaesthesiol. 2021 Oct 1;38(10):1042-1051. doi: 10.1097/EJA.0000000000001580. PMID 34366425
- [Derived] Li H, Guo J, Wang K, Zhang NR, Zheng ZN, Jin SQ. [Effect of open-lung ventilation strategy on oxygenation-impairment during laparoscopic colorectal cancer resection]. Zhonghua Wei Chang Wai Ke Za Zhi. 2020 Nov 25;23(11):1081-1087. doi: 10.3760/cma.j.issn.441530-20191209-00507. Chinese. PMID 33212557

DOCUMENTS (2):
  • Statistical Analysis Plan: statistical analysis plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03160144/SAP_001.pdf
  • Statistical Analysis Plan: Supplementary notes to the statistical analysis plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03160144/SAP_002.pdf